CLINICAL TRIAL: NCT03785015
Title: When Should Low-dose Aspirin be Resumed After Peptic Ulcer Bleeding? A Randomized Controlled Trial
Brief Title: When Should Low-dose Aspirin be Resumed After Peptic Ulcer Bleeding?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Beijing Friendship Hospital (Other); National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ReASA
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-06

CONDITIONS: Aspirin; GastroIntestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Withold aspirin till after endoscopic haemostasis (Experimental): Withhold the standard treatment of aspirin within 12 hours after endoscopic haemostasis.
  Interventions: Other: Resume Aspirin within 12 hours
- Withold aspirin till 72 hours (Active Comparator): Withhold the standard treatment of aspirin till 72 after endoscopic haemostasis.
  Interventions: Other: Resume Aspirin 72 - 84 hours

INTERVENTIONS:
Other: Resume Aspirin within 12 hours — Resume the standard treatment within 12 hours after endoscopic haemostasis
  Arms: Withold aspirin till after endoscopic haemostasis
Other: Resume Aspirin 72 - 84 hours — Resume the standard treatment between 72 and 84 hours after endoscopic haemostasis
  Arms: Withold aspirin till 72 hours

SUMMARY:
Acute upper gastrointestinal (GI) bleeding associated with the use of low-dose aspirin (ASA) is a major cause of peptic ulcer bleeding worldwide. Among survivors of acute myocardial infarction, a study of over 14,000 patients reported that the risk of life-threatening GI bleeding in the first two months is 7 times higher than that in the subsequent months. After endoscopic control of ulcer bleeding, most patients with cardiovascular (CV) diseases will need to resume ASA. However, the investigator found that immediate resumption of ASA saves life but at the expense of higher risk of recurrent bleeding. Peptic ulcer bleeding associated with ASA is a major cause of hospitalization in Hong Kong. Currently, ASA use has contributed to about one-third of the bleeding ulcers admitted to our hospital that serves a local population of 1.5 million. Accordingly, current international guidelines recommend early resumption of ASA but the optimal timing is unknown. Clinicians often face the dilemma: when should ASA be resumed? Furthermore, patients who suffer from acute peptic ulcer bleeding are often elderly patients with significant co-morbidities. Mortality in these patients remains high. Clinicians are facing an increasing number of patients who are on antiplatelet drugs or anticoagulants. The investigator proposes a open-label randomized-controlled trial to evaluate the optimal timing of resuming ASA in patients with CV diseases complicated by peptic ulcer bleeding. Patients will be randomized to resume the standard treatment within first few hours or only to resume the standard treatment 72 hours after endoscopic haemostasis.

DETAILED DESCRIPTION:
Acute upper gastrointestinal (GI) bleeding associated with the use of low-dose aspirin (ASA) is a major cause of peptic ulcer bleeding worldwide. Among survivors of acute myocardial infarction, a study of over 14,000 patients reported that the risk of life-threatening GI bleeding in the first two months is 7 times higher than that in the subsequent months (1). After endoscopic control of ulcer bleeding, most patients with cardiovascular (CV) diseases will need to resume ASA. Clinicians often face the dilemma: when should ASA be resumed? Furthermore, patients who suffer from acute peptic ulcer bleeding are often elderly patients with significant co-morbidities. Mortality in these patients remains high. Clinicians are facing an increasing number of patients who are on antiplatelet drugs or anticoagulants.

However, there are very limited data to guide the best timing for resumption of ASA in these high risk patients. To date, our group has conducted the only randomized controlled trial in the literature that has partially addressed this issue. Importantly, the investigator found that immediate resumption of ASA saves life but at the expense of higher risk of recurrent bleeding (2). Accordingly, current international guidelines recommend early resumption of ASA but the optimal timing is unknown.

In the setting of acute GI bleeding, it is often a dilemma whether to stop or to restart these drugs. The balance between bleeding and thrombotic risks is difficult and treatment is often empirical and not evidence-based.

The investigator aims to test the hypothesis that in ASA users complicated by peptic ulcer bleeding, withholding ASA till day 3 reduces the risk of recurrent bleeding compared to immediate resumption of ASA without a significant increase in mortality.

References

1. Moukarbel GV, Signorovitch JE, Pfeffer MA et al. Gastrointestinal bleeding in high risk survivors of myocardial infarction: the VALIANT Trial. Eur Heart J 2009;30(18):2226-32.
2. Sung JJ, Lau JY, Ching JY et al. Continuation of low-dose aspirin therapy in peptic ulcer bleeding: a randomized trial. Ann Intern Med 2010;152(1):1-9.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Patients with actively bleeding gastroduodenal lesions (peptic ulcer, bleeding erosions, or Dieulafoy's lesion) or ulcers showing other high risk stigmata (visible blood vessels or adherent clots) treated by endoscopic therapy
3. Subjects continue to require regular ASA or dual anti-platelet therapy for treatment of CV or cerebrovascular diseases after this bleeding episode

Exclusion Criteria:

1. Patients who received ASA for primary prophylaxis
2. Unsuccessful endoscopic hemostasis of bleeding ulcers or ulcer perforation
3. Gastric outlet obstruction
4. Known sensitivity to PPIs
5. Previous partial gastrectomy or vagotomy
6. Patients need concomitant anticoagulant
7. Pregnant unless sterilization, menopause or last menstrual period within 7 days
8. Other co-morbidities or advanced age that will hinder the drug compliance or follow up
9. Malignancy on active treatment
10. Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrent peptic ulcer bleeding | 30 days after endoscopic treatment
  Recurrent peptic ulcer bleeding within 30 days of endoscopic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Siew C Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No